CLINICAL TRIAL: NCT00223535
Title: Cognitive Remediation and Social Skills Training in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012-0013-164
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenia; Schizoaffective
Keywords: Schizophrenia; Cognitive Remediation; Social Skills Training; Psychosocial
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Remediation

INTERVENTIONS:
Behavioral: Cognitive Remediation
Behavioral: Social Skills Training

SUMMARY:
The purpose of this study is to examine whether patients who participate in cognitive remediation prior to a skills training program learn and perform the skills better than patients who do not participate in cognitive remediation.

DETAILED DESCRIPTION:
Subjects are 40 stable outpatients with schizophrenia or schizoaffective disorder who are receiving medication and routine follow-up care at community clinics in San Antonio, Texas.

Patients receive baseline assessments and then are randomly assigned to either Cognitive Remediation (CR) or Keyboarding Skills (KS) for a period of 8 weeks. Following 8 weeks of treatment in either CR or KS, all patients participated in Social Skills Training (SST) for a period of 8 weeks. Assessments conducted by raters blinded to treatment condition are repeated following either remediation or control treatment, and again following SST.

Treatment groups Cognitive Remediation (CR) -- The CR program is based upon teaching techniques developed within educational psychology that promote intrinsic motivation and task engagement. The program uses existing computer software packages (e.g., Oregon Trail) with engaging story lines or activities, and built-in reinforcement of correct responses to help patients with schizophrenia develop attention, memory, planning, and problem-solving skills. CR is delivered in a computer lab setting with a facilitator present to assist patients.

Keyboarding Skills (KS) -- Control Treatment: The control treatment is an engaging self-paced software program designed to teach typing skills. KS is delivered in a computer lab setting with a facilitator present.

Both the KS and CR are administered in small groups of three to five patients each.

Social Skills Training (SST) -- SST is a manual-driven, behavioral rehabilitation program teaching basic conversation and social problem-solving skills (Bellack et al., 1997). SST runs for 8 weeks and is conducted in small groups that meet twice weekly.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia/schizoaffective disorder
* currently receiving treatment with an atypical antipsychotic medication
* between the ages of 18 and 60 years
* speak English as their primary language
* has at least a 6th grade level of reading (WRAT) Exclusion Criteria
* no current diagnosis of substance abuse or dependence
* no documented history of head injury, epilepsy or mental retardation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2003-02; Study Completion 2005-03

PRIMARY OUTCOMES:
Scores on tests of cognitive functioning

SECONDARY OUTCOMES:
Outcomes on tests of social functioning after SST

CONTACTS AND LOCATIONS:
Overall Officials: Dawn I Velligan, Ph.D., Principal Investigator — University of Texas
Locations (1):
- UTHSCSA, San Antonio, Texas, United States